CLINICAL TRIAL: NCT05033158
Title: Investigation to Reveal the Immune Reaction Upon COVID-19 Vaccination in the Belgian Cancer Population: COVID-19 Protection and Vaccine Safety (REAL-V)
Brief Title: The Immune Reaction Upon COVID-19 Vaccination in the Belgian Cancer Population.
Acronym: REAL-V
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Antwerp (Other)
Collaborators: KomOpTegenKanker (non-profit organization) (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 001752
Record Dates: First submitted 2021-04-02; First posted 2021-09-02 (Actual); Last update posted 2023-06-15 (Actual); Status verified 2023-06

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cancer patients (Other): Level of antibodies against SARS-CoV-2 will be measured in these patients
  Interventions: Other: Blood sampling

INTERVENTIONS:
Other: Blood sampling — Blood sampling before and after COVID-19 vaccination

SUMMARY:
This study investigates the immune response in the cancer population in Belgium being vaccinated with an approved vaccine types being authorized for use in Belgium. This question needs to be answered to make sure that this vulnerable population is properly protected against possible SARS-CoV-2 infection and that vaccine administration is safe.

DETAILED DESCRIPTION:
Rationale: Patients with cancer have an increased risk of adverse outcome of COVID-19 and should be at high prioritisation for vaccination against SARS-CoV-2. The COVID-19 vaccine trials have not included cancer patients as such, the efficacy and duration of immunity in patients with cancer are still unknown. Keeping in mind that cancer patients are often immunocompromised, the immune response upon vaccination needs further investigation.

The REAL-V is a prospective, multicenter cohort study. The humoral immunity response based on anti-SARS-CoV-2 IgG antibodies upon COVID-19 vaccination will be investigated in blood samples taken 4 months, 6 months and 12 months after (first) vaccine administration. Potential factors that affect immunity, will be recorded, such as type and stage of cancer, anti-cancer treatment, concomitant medication,..To investigate the safety of different COVID-19 vaccines, incidence and severity of systemic adverse events will be reported using an App based system answering questionnaires about specific vaccine related complaints.

ELIGIBILITY:
Inclusion Criteria:

* Age of 18 years or older
* Oncological or hematological malignancy or history of it
* Life expectancy > 3 months
* Ability to provide informed consent

Exclusion Criteria:

* Women who are pregnant or breastfeeding
* Immune deficiency not related to cancer or cancer treatment
* Allergy (multiple); to be determined by physician

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 402 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2023-06-13 (Actual)

PRIMARY OUTCOMES:
Immune response | 4 months
  The primary endpoint is the quantification of different anti-SARS-CoV-2 specific IgG antibodies 4 months after (first) vaccine administration. Antibody titers to the full Spike, S1, S2, RBD (receptor binding domain) and N (nucleocapsid) protein of SARS-CoV-2 will be measured quantitatively. For this measurement a multiplex SARS-CoV-2 immunoassay will be used.

SECONDARY OUTCOMES:
Duration of the immune response | 6 months
  To study the evolution and duration of the immune response after vaccination: using serological assays to analyze anti-RBD IgG titers 6 months after (first) vaccine administration.
Neutralizing capacity | 6 months
  To analyze the titer of neutralizing antibodies both 4 and 6 months after (first) vaccine administration
Efficacy of the immune response | 12 months
  This will be assessed by the SARS-Cov2 infection rate based on information collected through questionnaires on incidence of (PCR-confirmed) SARSCoV-2 infection within a time-frame of 12 months after the start of the study.
Vaccine safety | 12 months
  Safety will be reported in terms of incidence and severity of systemic adverse events (AEs) during a continuous App based reporting system or using a questionnaire 3 days after vaccine administration.

CONTACTS AND LOCATIONS:
Overall Officials: Marc Peeters, Prof. MD, Principal Investigator — University Hospital, Antwerp
Locations (8):
- Belgium (8):
  - University Hospital Antwerp, Edegem, Antwerp
  - AZ Klina, Brasschaat
  - AZ Sint Jan, Bruges
  - UZ Brussel, Brussels
  - AZ Sint Lucas, Ghent
  - UZ Gent, Ghent
  - AZ Groeninge, Kortrijk
  - AZ Nikolaas, Sint-Niklaas

IPD SHARING:
Plan to Share IPD: No